CLINICAL TRIAL: NCT04235296
Title: Evaluation of the Safety and Effectiveness of Mesenchymal Stem Cell Conditioned Medium-derived Pleiotropic Factor in Treating Residual Burn Wound
Brief Title: Mesenchymal Stem Cell Conditioned Medium-derived Pleiotropic Factor in Treating Residual Burn Wound
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiaobing Fu, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHIN-PLAGH-MP-03
Record Dates: First submitted 2020-01-17; First posted 2020-01-21 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Mesenchymal Stem Cell-derived Pleiotropic Factor in Treating Residual Burn Wound
MeSH Terms: interventions — Epidermal Growth Factor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): epidermal growth factor
  Interventions: Biological: epidermal growth factor
- experimental group (Experimental): mesenchymal stem cell conditioned medium-derived pleiotropic factor
  Interventions: Biological: mesenchymal stem cell conditioned medium-derived pleiotropic factor

INTERVENTIONS:
Biological: epidermal growth factor — Residual wounds from the same person were divided into control group and experimental group. The epidermal growth factor is used to control group. Then the foam wound dressing was selected to cover the residual wound, and the dressing was changed every 2 days.
  Arms: control group
Biological: mesenchymal stem cell conditioned medium-derived pleiotropic factor — Residual wounds from the same person were divided into control group and experimental group. The pleiotropic factor is used to control group. Then the foam wound dressing was selected to cover the residual wound, and the dressing was changed every 2 days.
  Arms: experimental group

SUMMARY:
Treatment of extensive deep burn residual wounds is a common problem in burn plastic surgery. Due to bacterial invasion, excessive maturation of granulation tissue, poor abrasion resistance of new epithelium, and coexistence of wound healing and dissolution can lead to delayed wound healing. Residual wounds rarely heal spontaneously and are prone to recurrence. Mesenchymal stem cells (MSC) boost tissue repair through paracrine. Many biological effectors, including IGF-1, vascular endothelial growth factor (VEGF), TGF-β1 have been found in MSC conditioned media (MSC-CM), and play a role in promoting tissue repair and regeneration.Our previous animal experiments have confirmed the role of MSC-CM in regulating wound inflammation, repairing damaged repair cells and promoting wound regeneration. In here, we will evaluate the safety and effectiveness of mesenchymal stem cell conditioned medium-derived pleiotropic factor in treating residual burn wound.

ELIGIBILITY:
Inclusion Criteria:

Patients with thermal burns are all residual wounds that have not healed after 1 month; The distance between adjacent residual wounds of the same patient is greater than 10cm; Patients signing informed consent -

Exclusion Criteria:

Patients with severe heart, lung, liver, kidney, blood and mental system diseases; Combined with diabetes, hypertension and malnutrition; Patients with shock, severe systemic infections, and pregnant or lactating women. -

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-17 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
wound healing rate | 2 months
  Original wound area minus unhealed wound area divided by original wound area

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobing Fu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- PLA Central Theater Air Force Hospital, Datong, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Need to contact the researcher and open sharing after the researcher's consent
Supporting Information: Study Protocol
Time Frame: One year after completion of the clinical trial
Access Criteria: One year after completion of clinical trials